CLINICAL TRIAL: NCT02150915
Title: Acute Effects of Acupuncture in the Response of the Median Neurodynamic Test: a Randomised, Double-blind, Non-inferiority Trial
Brief Title: Acute Effects of Acupuncture in the Response of the Median Neurodynamic Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuno Morais (Other)
Collaborators: Instituto Politécnico de Leiria (Other)
Responsible Party: Sponsor-Investigator, Nuno Morais, Master student in traditional chinese medicine, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNT-ACUP-2014
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Other Lesions of Median Nerve
Keywords: Acupoints; Acupuncture therapy; Median nerve; Biomechanics
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- new acupoint (Experimental): Subjets in this arm receive acupuncture therapy in a new acupoint (leopard spot needling technique)
  Interventions: Other: Acupuncture therapy (leopard spot needling technique)
- classical acupoint (Active Comparator): Subjects in this arm receive acupuncture therapy in a classical acupoint in the pericardial conduit (leopard spot needling technique)
  Interventions: Other: Acupuncture therapy (leopard spot needling technique)

INTERVENTIONS:
Other: Acupuncture therapy (leopard spot needling technique) — Comparison of the effects of a new or extraordinary acupoint versus a classical acupoint

SUMMARY:
The purpose of this study is to test whether the application of acupuncture alters the mechanical (range of elbow extension motion) and physiological (eg, intensity and onset of discomfort, tingling feeling and/or feeling of tension or restriction of movement) responses of the neurodynamic test of nerve median in asymptomatic individuals

DETAILED DESCRIPTION:
To understand the potential of acupuncture therapy in pain syndromes that involve changes of the mechanics and physiology of the peripheral nervous system

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years-old
* normal mobility in the joints of the upper quadrant

Exclusion Criteria:

* pathology that may impair nerve function (eg, diabetes)
* complaints over the past 3 months in the upper quadrant
* significant deformities in the upper quadrant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Elbow extension range of motion | immediately after the application of acupuncture
  Elbow extension range of motion during the median nerve neurodynamic test is measured by means of a smartphone (iPhone 4; app Compass (native); iOS 7.1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Henry J Greten, PhD, Principal Investigator — Universidade do Porto - Instituto de Ciências Biomédicas Abel Salazar
Locations (1):
- Instituto de Ciências Biomédicas Abel Salazar - Universidade do Porto, Porto, Porto District, Portugal

REFERENCES:
- [Derived] Morais N, Greten HJ, Santos MJ, Machado JP. Immediate effects of acupuncture on the mechanosensitivity of the median nerve: an exploratory randomised trial. Acupunct Med. 2018 Jun;36(3):132-138. doi: 10.1136/acupmed-2016-011357. Epub 2018 May 2. PMID 29720378